CLINICAL TRIAL: NCT04625335
Title: Effects of Prophylactic Massage Therapy on Pain Tolerance and Threshold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyle Knight (Other)
Responsible Party: Sponsor-Investigator, Kyle Knight, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 15-0650-P1H
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Pain
Keywords: massage therapy; pain tolerance; pain threshold
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Intervention First (Experimental): Adult, healthy volunteers will receive the intervention (prophylactic therapeutic massage) before completing the Cold Pressor Test. Following the crossover, these participants will then complete the Cold Pressor Test without prior massage.
  Interventions: Other: No Massage Protocol; Other: Prophylactic Therapeutic Massage
- Group 2: Intervention Last (Experimental): Adult, healthy volunteers will complete the Cold Pressor Test without prior massage. After crossover, they will receive the intervention (prophylactic therapeutic massage) before completing the Cold Pressor Test.
  Interventions: Other: No Massage Protocol; Other: Prophylactic Therapeutic Massage

INTERVENTIONS:
Other: No Massage Protocol — Participants did not receive therapeutic massage prior to completing the Cold Pressor Test.
Other: Prophylactic Therapeutic Massage — Participants received a 5 minute prophylactic therapeutic massage prior to completing the Cold Pressor Test. The massage was completed distally-to-proximally in the following order: superficial strokes to the entire forearm, deep strokes to the entire forearm, one-handed palmar kneading of the entire forearm with participant's forearm stabilized by the massager's the other hand, bilateral thumb kneading of the forearm in strips until the entire forearm was addressed, bilateral transverse thumb motions over palmar surface of the hand, single thumb kneading of thenar and hypothenar eminences simultaneously, bilateral thumb kneading to the dorsum of hand, deep stroking to the entire forearm, and superficial stroking to the entire forearm.

SUMMARY:
Therapeutic massage has been thought to reduce anxiety and increase relaxation in human patients.This study is meant to determine the immediate effects of therapeutic massage on pain tolerance and threshold.

DETAILED DESCRIPTION:
Patients participated in two trials of a pain stimulus test that measured pain threshold and pain tolerance. One trial was titled "Massage Protocol" and the other, "No-Massage Protocol." During the "Massage Protocol," they received a therapeutic massage to the forearm before participating in the pain stimulus test. During the "No-Massage Protocol" they did not receive a massage before participating in the pain stimulus test. Their pain threshold and tolerance for both trials were compared against each other. Each patient was randomized as to which protocol they participated in first.

ELIGIBILITY:
Inclusion Criteria:

-generally healthy

Exclusion Criteria:

* pregnant
* smoker
* cold allergy
* Raynaud's disease
* cryophobia

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2015-10-02 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Change in Pain Tolerance | Approximately 3 minutes
  Pain tolerance is measured as using the Cold Pressor Test. It is calculated as the amount of time elapsed between submersion of the hand in cold water and removal due to intolerance of the stimulus. Data will be reported as the change in pain tolerance between massage and no massage.
Change in Pain Threshold | Approximated 3 minutes
  Pain threshold is measured using the Cold Pressor Test. It is calculated as the amount of time elapsed between submersion of the hand in cold water and the first report of pain. Data will be reported as the change in pain threshold between massage and no massage.

CONTACTS AND LOCATIONS:
Overall Officials: Terry Malone, PT, EdD, Study Director — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferrell-Torry AT, Glick OJ. The use of therapeutic massage as a nursing intervention to modify anxiety and the perception of cancer pain. Cancer Nurs. 1993 Apr;16(2):93-101. PMID 8477405
- [Background] Cherkin DC, Eisenberg D, Sherman KJ, Barlow W, Kaptchuk TJ, Street J, Deyo RA. Randomized trial comparing traditional Chinese medical acupuncture, therapeutic massage, and self-care education for chronic low back pain. Arch Intern Med. 2001 Apr 23;161(8):1081-8. doi: 10.1001/archinte.161.8.1081. PMID 11322842
- [Background] Field T, Hernandez-Reif M, Taylor S, Quintino O, Burman I. Labor pain is reduced by massage therapy. J Psychosom Obstet Gynaecol. 1997 Dec;18(4):286-91. doi: 10.3109/01674829709080701. PMID 9443139
- [Background] Cherkin DC, Sherman KJ, Deyo RA, Shekelle PG. A review of the evidence for the effectiveness, safety, and cost of acupuncture, massage therapy, and spinal manipulation for back pain. Ann Intern Med. 2003 Jun 3;138(11):898-906. doi: 10.7326/0003-4819-138-11-200306030-00011. PMID 12779300
- [Background] Hernandez-Reif M, Field T, Krasnegor J, Theakston H. Lower back pain is reduced and range of motion increased after massage therapy. Int J Neurosci. 2001;106(3-4):131-45. doi: 10.3109/00207450109149744. PMID 11264915
- [Background] Preyde M. Effectiveness of massage therapy for subacute low-back pain: a randomized controlled trial. CMAJ. 2000 Jun 27;162(13):1815-20. PMID 10906914
- [Background] National Institute on Drug Abuse; Johns Hopkins University. Study of the treatment of experimental pain in opioid dependent persons on methadone or buprenorphine maintenance. In: ClinicalTrials.gov [Internet]. Bethesda (MD): National Library of Medicine (US). 2015-[cited 2015 Aug 19]. Available from: https://clinicaltrials.gov/ct2/show/NCT01642030 NLM Identifier: NCT01642030.
- [Background] Kelly D. Therapeutic massage of the forearm and hand. Lecture presented at: PT615 Basic Clinical Skills; 2015; University of Kentucky, Lexington, KY.